CLINICAL TRIAL: NCT06052475
Title: Physiological Versus Right Ventricular Outcome Trial Evaluated for Bradycardia Treatment Upgrades
Acronym: PROTECT-UP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23HH8156
Record Dates: First submitted 2023-09-19; First posted 2023-09-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pacing-Induced Cardiomyopathy; Heart Failure
Keywords: Physiological Pacing; RV Pacing; Biventricular Pacing; Pacemaker Upgrade
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiological Pacing (Conduction System Pacing or Biventricular Pacing) (Experimental): The approach for physiological pacing will be either His bundle pacing or left bundle pacing at the operator's discretion. If both of these are not achieved biventricular pacing will be performed.
  Interventions: Device: Physiological Pacing Upgrade (Conduction System Pacing or Biventricular Pacing)
- Right Ventricular Pacing (Active Comparator): Right ventricular pacing (apical or septal lead locations as per the implanting physicians' normal practice)
  Interventions: Device: Continued RV Pacing (Right Ventricular Pacing)

INTERVENTIONS:
Device: Physiological Pacing Upgrade (Conduction System Pacing or Biventricular Pacing) — The approach for physiological pacing upgrade will be either His bundle pacing or left bundle pacing at the operator's discretion. If both of these are not achieved biventricular pacing will be performed.
  Arms: Physiological Pacing (Conduction System Pacing or Biventricular Pacing)
Device: Continued RV Pacing (Right Ventricular Pacing) — Right ventricular pacing (apical or septal lead locations as per the implanting physicians' normal practice).
  Arms: Right Ventricular Pacing

SUMMARY:
Guidelines for patients having first-time implants advocate that even when heart function is only mildly impaired, modern pacing approaches should be utilised to avoid the potentially damaging effects of RV pacing to preventing symptoms from pacing induced or worsened cardiomyopathy.

However, once a traditional (RV) pacemaker is implanted, development of impaired heart function does not prompt a device upgrade. Even at the end of battery life, physicians simply replace it like-for-like.

This trial tests whether such patients have better symptoms and quality of life if changed to a modern physiological pacing strategy from the traditional RV pacing approach.

In this crossover trial, participants will be upgraded to a physiological pacing strategy.

After their procedure, they will have a one-month run-in period to recover from the procedure (their pacemaker will be programmed to continued RV pacing).

They will be have 2 one-month blinded time periods, randomised to physiological pacing or right ventricular pacing alternately. They will subsequently undergo two six-month blinded randomised time periods.

Patients will document symptoms monthly on a mobile phone application or computer. At the end of each time period, they will have measurements of heart function, a walking test and quality-of-life questionnaires including the SF-36 questionnaire.

The investigators hypothesise that upgrading to physiological pacing strategies will improve patients' quality of life.

ELIGIBILITY:
Patients with an RV pacemaker and LVEF 35-50% and a high burden of right ventricular pacing (>40%) who are clinically indicated for a cardiac resynchronisation therapy upgrade procedure and:

1. EF reduced by >5% of increase in LVESV by 10ml since implant
2. NT-proBNP >250ng/L in sinus rhythm
3. NT-proBNP > 750 Ng/L if AF
4. Left atrial volume index > 30ml/m2
5. Regular loop diuretics prescribed
6. Decline in daily patient activity by >1 hour per day since implant
7. Decrease in device measured thoracic impedance
8. Patient reported decline in functional class or exercise tolerance

Exclusion Criteria:

* Those unable to provide informed consent
* Patients under age 18
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
SF-36 (Short Form 36 Health Survey Questionnaire) Physical Component Summary | From date of baseline, until end of trial follow-up at fourteen months post-baseline

SECONDARY OUTCOMES:
Left ventricular ejection fraction | From date of baseline, until end of trial follow-up at fourteen months
  (% ejection fraction)
Left ventricular end systolic volume | From date of baseline, until end of trial follow-up at fourteen months
  (millilitres)
Minnesota Living with Heart Failure Questionnaire | From date of baseline, until end of trial follow-up at fourteen months
Six-minute walk test | From date of baseline, until end of trial follow-up at fourteen months
  Measured in distance in metres
Atrial fibrillation | From date of baseline, until end of trial follow-up at fourteen months
  (atrial fibrillation percentage burden as measured by pacemaker device - %)
Patient preference based on blinded symptomatic preference | At 2 months following baseline and 14 months following baseline visit
EQ-5D Questionnaire | From date of baseline, until end of trial follow-up at fourteen months post-baseline visit
  EQ-5D is the name of the instrument and is not an acronym. The EQ-5D-5L consists of 2 pages: the EQ-5D descriptive system and the EQ 'visual analogue scale' (EQ VAS).
  The descriptive system is made up of 5 sections: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative (numerical) measure of health outcome that reflect the patient's own judgement. A high score on the VAS means a better outcome. A low score on the VAS means a worse outcome.
Patient symptoms assessed on a scale of 0-100 monthly | From date of baseline, until end of trial follow-up at fourteen months post-baseline visit
  This questionnaire will be sent to participants on a monthly basis for the duration of the study
Safety endpoints | From device implant date, assessed up to 15 months at the end of the trial (including a one-month run-in period post-procedure prior to the first baseline visit)
  Device infections (requiring device extraction), pacing thresholds, need for lead revision or reimplantation, generator change, haematoma and pneumothorax
SF-36 (Short Form 36 Health Survey Questionnaire) Overall Score | From date of baseline, until end of trial follow-up at fourteen months post baseline visit
SF-36 (Short Form 36 Health Survey Questionnaire) Individual Component Scores | From date of baseline, until end of trial follow-up at fourteen months post baseline visit
BNP (B-type natriuretic peptide) | From date of baseline, until end of trial follow-up at fourteen months post baseline visit
  B-type natriuretic peptide blood test

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Keene, PhD, Principal Investigator — Imperial College London; Nandita Kaza, MRCP, Study Director — Imperial College London; Matthew Shun-Shin, PhD, Study Director — Imperial College London
Locations (12):
- United Kingdom (12):
  - Royal Papworth Hospital, Cambridge
  - St. Richard's Hospital - University Hospitals Sussex, Chichester
  - University Hospitals Coventry and Warwickshire NHS Trust,, Coventry
  - Croydon University Hospital - Croydon Health Services, Croydon
  - Glenfield Hospital, Leicester
  - Hammersmith Hospital, London
  - King's College Hospital, London
  - St Bartholomew's Hospital - Barts Health NHS Trust, London
  - Oxford University Hospitals, Oxford
  - University Hospitals Southampton, Southampton
  - Great Western Hospitals, Swindon
  - Worthing Hospital - University Hospitals Sussex, Worthing

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-29): https://cdn.clinicaltrials.gov/large-docs/75/NCT06052475/Prot_SAP_002.pdf